CLINICAL TRIAL: NCT06492083
Title: A Randomized Controlled Clinical Stuty on the Treatment and Nursing Care of CIPN Patients With Traditional Chinese Medicine Hot Package
Brief Title: A Stuty on the Treatment and Nursing Care of CIPN Patients With Traditional Chinese Medicine Hot Package
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KY-2024-076
Record Dates: First submitted 2024-06-18; First posted 2024-07-09 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy
Keywords: Chemotherapy-Induced Peripheral Neuropathy/CIPN; hot compress with chinese herbal packets

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): All chemotherapies were strictly followed by drug-use routine. The paclitaxel and platinum administration rate were set as 180ml/h. Health guidance should provide before and after chemotherapies, including precautions for chemotherapy, dietary guidance, life guidance, etc. For patients with peripheral neuropathy that gradually worsen and affect muscle and joint functions, environmental management and self-management should be guided to prevent from falls, bumps, scalds, frostbite, sharps and other accidents.
- observation group (Experimental): In addition to the usual nursing measures of the control group, traditional Chinese medicine was used for acupoint treatment and home care：Patients are consulted by TCM specialist nurses and join the WeChat group to complete the hot package home care health education. Heat herbal packets and keep the temperature at 40-50 °C, fix the hot bag on the corresponding acupuncture points of each limb for 30 minutes. Chemotherapy should not be used on the same day and the next day, and the rest of the time should be treated with hot package every day.
  Interventions: Other: traditional Chinese medicine hot bag

INTERVENTIONS:
Other: traditional Chinese medicine hot bag — traditional Chinese medicine hot bag
  Arms: observation group

SUMMARY:
The combination of platinum and taxane drugs has a chemotherapy-induced peripheral neuropathy (CIPN) rate of 73% to 83%. Its symptoms can not only limit daily activities and cause a variety of accidental injuries, but also easily cause negative emotions and seriously affect the quality of life. Modern Western medicine lacks effective clinical intervention methods, and the treatment of acupuncture points with traditional Chinese medicine is simple to operate, easy to observe adverse reactions, and is suitable for continuous self-treatment outside the hospital after training, saving patients time to travel to and from the hospital, and high patient acceptance. Due to the similarity of the pathogenesis of some traditional Chinese and Western medicine in CIPN and the effectiveness of its application in patients with DPN, this study evaluated the effect of specific formulations of Chinese medicine on CIPN by comparing the degree of nerve damage between the following formulations of Chinese medicine hot packs in patients with platinum combined with paclitaxel chemotherapy and the control group.

DETAILED DESCRIPTION:
A random group generator was used to divide the sample of 90 cases, and 45 cases in the control group and 45 cases in the intervention group.

Control group: The chemotherapy was strictly followed by the drug use routine, administered by central vein, paclitaxel and platinum administration rate were set at 180ml/h, and routine health guidance was given before and after chemotherapy.

Intervention group: In addition to the usual nursing measures of the control group, traditional Chinese medicine hot bao acupoint treatment and home care were used.

Patients in both the intervention and control groups were assessed for peripheral neuropathy on the 14th day after the completion of each two rounds of chemotherapy, and the NCI-CTCAE, FACT/GOG-Ntx, and KPSS score scales were assigned according to the patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult and kinetic patients expected survive with tumor for more than 1 year. Those who use platinum in combination with paclitaxel for chemotherapy for the first time; Voluntarily agree to participate and sign a consent form

Exclusion Criteria:

* Those who are allergic to platinum, paclitaxel or Chinese herbal medicine ingredients; Patients with diabetes mellitus, Raynaud's syndrome, central or peripheral nerve disease symptoms; Those who cannot judge their own symptoms; Pregnant / lactating women; Patients with advanced rheumatoid arthritis, severe joint deformity or incapacitation; Those with other immune system diseases； Patients who have not completed the chemotherapy regimen; Patients who were not treated with hot acupuncture points as prescribed (missed dosing ≥ 3 times per week); Incomplete collection of clinical data; Subjects who voluntarily request to withdraw from this treatment, or are unwilling to continue treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Sensory neuropathy | 6 months
  National Cancer Institute-Common Terminology Criteria for Adverse Events. Scoring form 1 to 5 degree.
Motor neuropathy Motor neuropathy | 6 months
  National Cancer Institute-Common Terminology Criteria for Adverse Events. Scoring from 1 to 5 degree.

SECONDARY OUTCOMES:
Numbness, tingling sensation or comfortlessness in the limbs | 6 months
  Functional assessment of cancer therapy /gynaecologic oncology group-neuro-toxicity.Scoring from 0 to 4.
Joint muscle pain | 6 months
  Functional assessment of cancer therapy /gynaecologic oncology group-neuro-toxicity.Scoring from 0 to 4.
Hearing difficulties Hearing difficulties or tinnitus | 6 months
  Functional assessment of cancer therapy /gynaecologic oncology group-neuro-toxicity.Scoring from 0 to 4.
Pace impairment | 6 months
  Functional assessment of cancer therapy /gynaecologic oncology group-neuro-toxicity.Scoring from 0 to 4.
Sense of small objects | 6 months
  Functional assessment of cancer therapy /gynaecologic oncology group-neuro-toxicity.Scoring from 0 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Dong, Bachelor, Principal Investigator — The Fourth Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- the Fourth Affiliated Hospital of School of Medicine, and International School of Medicine, International Institutes of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No